CLINICAL TRIAL: NCT04437225
Title: Renal Metabolism of Glycolate to Oxalate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sonia Fargue, Principle Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB160505004-GLI; K01DK114332 (NIH); UAB (Other: UAB)
Record Dates: First submitted 2020-06-15; First posted 2020-06-18 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Healthy
Keywords: oxalate metabolism; kidney stones; glycolate; isotope tracer study; urolithiasis; oxalate
MeSH Terms: conditions — Kidney Calculi; Urolithiasis

STUDY DESIGN:
Intervention Model Description: Subject will undergo the gold-standard technique of steady-state intravenous infusion of 13-glycolate administration. Selected subjects will also undergo other modified modalities of 13-glycolate administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Constant Infusion of 13C2-Glycolate (Experimental): Subjects will consume a controlled diet for 5 days total. On Days 3 and 4, subjects will collect 24 hour urines. On Day 5, they will come to the Clinical Research Unit (CRU) in the fasted state for a visit lasting from 7:00 am to 5:30 pm. An intravenous (IV) catheter will be placed in a vein on the back of the hand at 7:30 am for the carbon 13 glycolate infusion which will occur at a constant rate for 10 hours, following a priming dose. From 7:30 am to 5:30 pm, urine collections will occur hourly, and from 8:30 am to 5:30 pm, IV blood collections will occur every half hour. Subjects will receive a meal at 5:30 pm, thus concluding the CRU visit. At home, subjects will collect timed urine until the next morning to be returned to the CRU.
  Interventions: Dietary Supplement: Low oxalate controlled Diet; Other: Primed, continuous intravenous infusion of 13C2-Glycolate
- Single Intravenous Dose of 13C2-Glycolate (Experimental): Subjects will consume a controlled diet for 5 days total. On Days 3 and 4, subjects will collect 24 hour urines. On Day 5, they will come to the Clinical Research Unit (CRU) in the fasted state for a visit lasting from 7:00 am to 2:30 pm. An intravenous (IV) catheter will be placed in a vein on the back of the hand at 8:30 am for a single dose of carbon-13 glycolate to be administered. From 7:30 am to 2:30 pm, urine collections will occur hourly. At 8:30 am, IV blood samples will be taken every fifteen minutes until 9:30 am, every half hour from 9:30 am to 10:30 am, and then finally hourly from 10:30 am to 2:30 pm . Subjects will receive a meal at 2:30 pm, thus concluding the CRU visit. At home, subjects will collect timed urine until the next morning to be returned to the CRU.
  Interventions: Dietary Supplement: Low oxalate controlled Diet; Other: Bolus intravenous infusion of 13C2-Glycolate
- Single Oral Dose of 13C2-Glycolate (Experimental): Subjects will consume a controlled diet for 5 days total. On Days 3 and 4, subjects will collect 24 hour urines. On Day 5, they will come to the Clinical Research Unit (CRU) in the fasted state for a visit lasting from 7:00 am to 2:30 pm. At 8:30 am, subjects will ingest the carbon-13 glycolate, dissolved in to 50 ml (about 1/4 cup) of water. From 7:30 am to 2:30 pm, urine collections will occur hourly. At 8:30 am, intravenous (IV) blood samples will be taken every fifteen minutes until 9:30 am, every half hour from 9:30 am to 10:30 am, and then finally hourly from 10:30 am to 2:30 pm . Subjects will receive a meal at 2:30 pm, thus concluding the CRU visit. At home, subjects will collect timed urine until the next morning to be returned to the CRU.
  Interventions: Dietary Supplement: Low oxalate controlled Diet; Other: Oral bolus administration of 13C2-Glycolate

INTERVENTIONS:
Dietary Supplement: Low oxalate controlled Diet — Participants will consume a diet that is controlled in its contents of protein, carbohydrates, fat, calcium, oxalate, vitamin C and sodium. Participants will be asked not to take any dietary supplements, exercise strenuously, or consume food or drink that is not provided to them.
Other: Primed, continuous intravenous infusion of 13C2-Glycolate — Participants will receive a continuous intravenous administration of carbon-13 glycolate, a naturally occurring form of glycolate, over the course of several hours until steady-state is achieved, using an IV catheter.
  Other Names: Constant infusion of 13C2-Glycolate
  Arms: Constant Infusion of 13C2-Glycolate
Other: Bolus intravenous infusion of 13C2-Glycolate — Participants will receive a bolus intravenous administration of carbon-13 glycolate, a naturally occurring form of glycolate, using an IV catheter.
  Other Names: Single intravenous dose of 13C2-Glycolate
  Arms: Single Intravenous Dose of 13C2-Glycolate
Other: Oral bolus administration of 13C2-Glycolate — Participants will orally ingest a single dose of carbon-13 glycolate, a naturally occurring form of glycolate.
  Other Names: Single oral dose of 13C2-Glycolate
  Arms: Single Oral Dose of 13C2-Glycolate

SUMMARY:
This study will determine the contribution of glycolate metabolism to urinary oxalate excretion in healthy subjects, using carbon 13 isotope glycolate tracer technique and a low-oxalate controlled diet.

DETAILED DESCRIPTION:
It is known that glycolate, an intermediary molecule in normal metabolism, can be converted into oxalate. The origin of urinary oxalate is of interest as calcium oxalate is a main component of kidney stones. In the rare disease primary hyperoxaluria, excessive production of oxalate by the body results in frequent kidney stones and can cause loss of kidney function. Primary hyperoxaluria is caused by deficiencies in one of several enzymes involved in the glycolate pathway.

This study will seek to determine how much oxalate is formed from glycolate in normal subjects. After consuming a controlled diet, subjects will either ingest or have an intravenous infusion of carbon 13 glycolate, a stable isotope of glycolate that can be tracked and will also label downstream metabolic products. Blood and urine samples will be assessed for their amounts of labeled glycolate and labeled oxalate to provide an accurate measure of how much oxalate is made from normal glycolate breakdown in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent adults, able to read and comprehend the consent form
* 18-75 years of age
* Body Mass Index (BMI) between 19 and 40
* In good health as judged from a medical history, reported medications, and a complete blood metabolic profile
* Acceptable 24 hour urine collections (performed twice for screening)

Exclusion Criteria:

* History of any hepatic, renal, bowel, or endocrine disease or any other condition that may influence the absorption, transport or urine excretion of ions
* Abnormal urine chemistries or blood metabolic profiles
* Poor 24 hour urine collections completed during screening, judged by 24 hour urine creatinine excretion (indicative of not collecting all urine in the 24 hour period)
* Pregnancy, intention to become pregnant in the near future, or lactation
* Aged <18 or >75
* BMI <19 or >40

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Urinary oxalate measured by ion chromatography coupled with mass spectrometry | day 5 of dietary control
  Measurement of carbon 13 labeled and unlabeled urinary oxalate following carbon 13 glycolate administration, after equilibration under a low-oxalate diet.
Plasma glycolate measured by ion chromatography coupled with mass spectrometry | day 5 of dietary control
  Measurement of carbon 13 labeled and unlabeled plasma glycolate following carbon 13 glycolate administration, after equilibration under a low-oxalate diet.

SECONDARY OUTCOMES:
Urinary creatinine | day 5 of dietary control
  Baseline assessment of 24hr urinary creatinine under controlled low-oxalate diet.
Urinary glycolate measured by ion chromatography coupled with mass spectrometry | day 5 of dietary control
  Measurement of carbon 13 labeled and unlabeled urinary glycolate following carbon 13 glycolate administration, after equilibration under a low-oxalate diet.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Fargue, M.D., Ph.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States